CLINICAL TRIAL: NCT05014022
Title: Non-recovery of Kidney Function After AKI: Identifying High Risk Groups and Assessment With Multiparametric Renal MRI
Brief Title: Non-recovery of Kidney Function After AKI
Acronym: RECOVER-AKI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 21057; 302569 (Other: IRAS)
Record Dates: First submitted 2021-08-04; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples will be collected and frozen for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multiparametric renal MRI — 10 patients in the cohort will undergo MRI scanning at day 30 and 90

SUMMARY:
One in five patients admitted to hospital suffer a sudden reduction in kidney function, termed acute kidney injury (AKI). Rather than kidney 'injury' being caused by physical trauma, the term describes reversible damage caused by conditions such as being dehydrated or having an infection. Having AKI puts patients at an increased risk of long-term health problems, especially chronic kidney disease (CKD). CKD can also lead to other important health problems including a higher risk of heart disease and stroke. If we can reduce the progression of AKI to CKD this will benefit patients.

Currently, there is a gap in the follow-up of patients after AKI due to a lack of evidence about which patients should be followed up and when. Treatments for AKI during the episode and afterwards to prevent CKD are limited. This is mainly due to a lack of understanding about how and when the kidney recovers after AKI. New tools are needed in order to better identify patients at risk of CKD after AKI. This study aims to address these gaps in our knowledge by studying a group of AKI patients in detail.

Ultimately, the aim of this study is to produce results that will allow better planning of follow-up for patients as well the planning of future research to develop new treatments to reduce the risk of CKD in people recovering from AKI.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a sudden loss of renal function occurring in up to 20% of hospitalised patient. People who survive an episode of AKI are at increased risk of long-term effects on their health, in particular the development or progression of chronic kidney disease (CKD). At present, there are no interventions proven to reduce the development of CKD after an episode of AKI.

A significant gap exists in the current provision of post-AKI follow-up care. Current methods of assessing renal recovery are overly reliant on serum creatinine, an imperfect measure that over-estimate the degree of renal recovery due to the effect of critical illness on muscle mass. Based on expert opinion only, it is currently recommended that everyone who has experienced AKI should have kidney function and albuminuria checked at 90 days. In reality, current practice falls significantly below these standards. Less than half of patients with the most severe AKI see a nephrologist after discharge. Even for patients who have required dialysis for AKI, follow-up rates can be as low as 12%. Lack of evidence prevents a more evolved approach. Improving post-AKI care and reducing the development or progression of CKD could therefore directly benefit large numbers of patients. This is particularly pertinent with the additional restrictions on hospital appointments due to COVID-19. More evidence is urgently needed to inform which patients need follow-up and to integrate new techniques that significantly improve assessments of renal recovery.

Important knowledge gaps make it difficult to move directly to testing new interventions in randomised trials. AKI is not a single condition, rather a heterogeneous syndrome with a variety of causes affecting a wide range of people. Outcomes differ between clinical settings and are affected by factors related to AKI (e.g. its severity or duration), but also by an individual's co-existing long-term conditions, and possibly by their frailty. As well as CKD development, AKI is associated with higher long-term mortality rates, increased heart failure events, hospital readmissions, recurrent AKI and poorer quality of life. Which groups are most at risk of the different outcomes is not well established; similarly the groups that would have the greatest benefit from interventions to reduce the development of CKD are not currently known. It is therefore likely that subgroups of people who have sustained AKI will benefit from different models of post- AKI care i.e. a one-size fits all approach is unlikely to be beneficial or cost-effective. Finally, the timing of the renal recovery phase after an episode of AKI is poorly understood outside of experimental models, which differ in a number of ways from clinical AKI. Failure of recovery of creatinine by 90 days after AKI strongly associates with subsequent long-term reductions in renal function, suggesting that interventions may be needed prior to this time point, but descriptions of renal recovery between AKI and 90 days are lacking.

MRI has emerged as an imaging modality with promise to improve the understanding and characterisation of renal pathophysiology. It is a versatile technique in which structural and functional MRI measurements can be performed in a single multiparametric scan session to assess altered renal tissue microstructure, oxygenation, perfusion and blood flow. MRI is non-invasive, safe and avoids sampling bias by characterising the entire kidney with high spatial resolution. MRI does not involve ionising radiation, is repeatable (allowing serial assessments over time) and the MRI measures do not require gadolinium contrast agents. A series of recent systematic reviews covering the main functional renal MRI measures conclude that evidence is now needed to accelerate the translation of multiparametric renal MRI for clinical use. The reviews focussed on: arterial spin labelling (ASL, a measure of renal perfusion); Blood Oxygen Level Dependent (BOLD, sensitive to changes in renal oxygenation); longitudinal (T1) relaxation time (increases with scarring, correlates with fibrosis in the heart and liver; diffusion weighted imaging (DWI, sensitive to changes in renal tissue microstructure); and Phase Contrast (PC-MRI, a measure of renal artery blood flow).

Considering the high incidence of AKI, the long-term consequences of AKI present a major unmet clinical need affecting large numbers of people, with no proven interventions nor data to inform optimal care provision. If patients at risk of developing CKD could be better identified, this would provide a basis upon which interventions to improve patient outcomes could be planned.

The outputs of this study would directly inform planning of future research in the following ways:

* Collection of data supporting a larger prospective cohort study of AKI patients, using data from this study to directly inform study design and MRI protocols
* Identification of those at greatest risk of developing CKD after AKI will make clinical trials more efficient and more likely to succeed
* Increasing understanding of the time course of renal recovery will allow planning of the optimal time points for interventions and patient follow-up
* Demonstrate the potential application of renal MRI in NHS scanners leading to improved clinical evaluation of patients

ELIGIBILITY:
Inclusion Criteria:

* ≥18yrs
* Acute kidney injury stage 1-3 by KDIGO criteria
* At least one previous serum creatinine result available for determining baseline renal function
* Able to give informed consent

Exclusion Criteria:

* Unable to give consent or understand written information
* Obstructive uropathy
* Renal transplant
* Patient receiving palliative care
* Patient with AKI due to recent nephrectomy
* Patients with known or suspected acute vasculitis or glomerulonephritis requiring immunosuppression
* End-stage kidney disease (CKD stage G5 or already on RRT)
* Serum creatinine changes that do not meet the KDIGO definition of AKI

MRI cohort:

* Contraindications to MRI e.g. claustrophobia, cardiac pacemaker, metallic fragments or implants
* Age < 50years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital inpatients at Royal Derby Hospital across all areas.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who have non-recovery of renal function after an episode of AKI | 30, 60 and 90 days
  Defined as improvement of creatinine to less than 50% above baseline i.e. reversal of AKI diagnostic criteria

SECONDARY OUTCOMES:
90 day mortality | 90 days
  Day 90 data - based on status (alive/dead) at day 90
Hospital readmission rates | 90 days
  Number of times patients has been admitted to hospital based on hospital records
Quality of life score | 90 days
  Based on EQ5D (euroqol.org) scoring system. Descriptive scoring, lower number = higher quality of life
Fatigue score | 90 days
  Based on Brief Fatigue Inventory scoring (lower score = less fatigue)
Number of patients who have ongoing albuminuria over time | Day 30,60 and 90
  Progression / recovery over time. Urine albumin:creatinine ratio
Descriptive analysis of preferred follow-up models | 90 days
  Based on structured questioning of participants
Change in renal structure over time | Day 30 & 90
  As measured by T1, total kidney volume & DWI
Change in renal haemodynamics over time | Day 30 & 90
  As measured by ASL and phase-contrast MRI
Change in renal oxygenation over time | Day 30 & 90
  As measured by TRUST MRI